CLINICAL TRIAL: NCT02887144
Title: Investigating the Safety and Performance of SenSura Test Product in Subjects With Ileostomy
Acronym: CP257
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Coloplast - CP257
Record Dates: First submitted 2015-12-17; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura test product 1pc (Experimental): Subjects randomized to treatment sequence 1test:
  1. SenSura test product
  2. SenSura
  Interventions: Device: SenSura; Device: SenSura test product
- SenSura 1pc (Experimental): Subjects randomized to treatment sequence 2 test:
  1. SenSura
  2. SunSura test product
  Interventions: Device: SenSura; Device: SenSura test product

INTERVENTIONS:
Device: SenSura — SenSura is a Commercial and CE-marked ostomy product (1pc) manufactured by Coloplast A/S
Device: SenSura test product — SenSura test product is a CE-marked ostomy product (1pc) manufactured by Coloplast A/S

SUMMARY:
The aim of the current Investigation is to evaluate the safety and performance of SenSura test product 1pc flat and convex light compared with commercial SenSura.

DETAILED DESCRIPTION:
Investigators want to measure degree of leakage on a 4-point scale of SenSura and SenSura test product.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Be able to handle the products themselves
4. Have an ileostomy (end or loop ostomy) with a diameter between 10 - 40 mm
5. Have had their ileostomy for at least 3 months
6. Have used a 1-piece flat or convex light ostomy appliance with an open bag within the last month
7. Currently using midi or maxi bags
8. Willing to use minimum 1 product every second day (max. 2 days wear time)
9. Be mentally and physically capable of understanding and following the study procedures and completing the Case Report Form
10. Must be able to cut products themselves

Exclusion Criteria:

1. Currently receiving or have received within the past 2 months chemo- or/and radiation therapy
2. Currently receiving or have received within the past month local or systemic steroid treatment in the peristomal area
3. Are pregnant or breastfeeding
4. Participating in other interventional clinical investigations or have previously participated in this investigation
5. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin).
6. Known hypersensitivity of the product components and/or ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Degree of leakage | patients will test the products for 4 weeks
  Leakage under and outside the baseplate will be assessed by a 4 point leakage scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No